CLINICAL TRIAL: NCT07370584
Title: A Randomized, Vehicle-Controlled, Double-Masked Study of the Safety of IVMED-85 Ophthalmic Solution in Healthy Adults
Brief Title: A Safety Study of IVMED-85 Ophthalmic Solution in Healthy Adults
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: iVeena Delivery Systems, Inc. (Industry)
Collaborators: Lexitas Pharma Services, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IVNA 22-02
Record Dates: First submitted 2026-01-19; First posted 2026-01-27 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Safety Study
Keywords: eye drops; safety; myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vehicle ophthalmic solution (Placebo Comparator): Vehicle ophthalmic solution, administered twice a day
  Interventions: Drug: Vehicle Ophthalmic Solution
- IVMED-85 ophthalmic solution (Experimental): IVMED-85 ophthalmic solution (0.20 mg/mL)
  Interventions: Drug: IVMED-85 ophthalmic solution

INTERVENTIONS:
Drug: IVMED-85 ophthalmic solution — IVMED-85 ophthalmic solution (0.20 mg/mL), administer twice a day (morning and evening) in both eyes
  Arms: IVMED-85 ophthalmic solution
Drug: Vehicle Ophthalmic Solution — Vehicle ophthalmic solution, administer twice a day (morning and evening) in both eyes
  Arms: Vehicle ophthalmic solution

SUMMARY:
The purpose of this trial is to determine the safety of IVMED-85 eye drops in healthy adult subjects. Participants will be assigned to either the active or vehicle eyedrop group. The participants will receive eye drops twice daily for 6 weeks. Participants will not know which eyedrop they are taking.

DETAILED DESCRIPTION:
Randomized, double-masked, controlled studies are the gold standard of clinical research. This is a randomized, vehicle-controlled, double-masked Phase 1 clinical study to assess the safety of IVMED-85 ophthalmic solution in healthy adult subjects. 36 subjects (ages 18-49) will be randomly and equally assigned to one of two treatment groups: vehicle ophthalmic solution or 0.20 mg/mL IVMED-85 ophthalmic solution.

All subjects will dose twice daily (BID), morning and evening, in both eyes for 6 weeks. Subjects will attend 3 clinic visits (screening/baseline, Day 21, and Day 42 at which safety will be assessed. If any treatment-related adverse events occur, additional visits to monitor for resolution and/or treatment, at the Investigator's discretion, with at least 1 such visit occurring months 3 after the last study visit.

In this study, the vehicle is the control treatment, chosen to help ensure that any effect observed in the IVMED-85 group is due to the active ingredient. IVMED-85 will be administered as an eye drop, a common route of administration.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who meet all the following inclusion criteria at Visit 1 will be eligible to enroll in the study. Ocular criteria apply to both eyes.

  1. Age 18-49. -
  2. Ability to voluntarily provide written informed consent. -
  3. Being clinically healthy, as determined by the investigator. -
  4. Willing and able to comply with clinic visits and study-related procedures. -
  5. Willing and able to discontinue use of topical ocular medications, unless approved by investigator. Note: Artificial tears are allowed but must not be used within 30 minutes before or after administration of the study investigational product (IP). -
  6. BCVA better than or equal to 0.2 logarithm of the minimum angle of resolution (logMAR) (20/30 Snellen equivalent). -
  7. Corneal thickness 450 to 670 μm. -
  8. Intraocular pressure (IOP) ≤22 mmHg. -
  9. Willingness to not wear mascara for 6 weeks of the study. -
  10. Willingness to not swim in an indoor pool for 6 weeks of the study. -

Exclusion Criteria:

Subjects who meet any of the following criteria at Visit 1 will not be eligible to enroll in the study. Ocular criteria apply to either eye.

1. Participation in a clinical trial with the use of any investigational drug or treatment within 30 days prior to Visit 1 and duration of the study. -
2. Known copper allergy, sensitivity, or processing disorder (e.g., Wilson's disease). -
3. Presence of significant central corneal scarring or hydrops. -
4. History or presence of punctal stenosis or bloody discharge. -
5. History of or presence of nasolacrimal duct occlusion, nasolacrimal system trauma, nasolacrimal or eyelid cancer, ectropion or entropion, dacryocystitis, dacryoadenitis, chronic conjunctivitis, recurrent subconjunctival hemorrhage, trichiasis, distichiasis, or uncontrolled dry eye. -
6. Previous cornea, glaucoma, eyelid, strabismus (exotropia or esotropia), or intraocular surgeries. -
7. Current or previous ocular disorder, including but not limited to: strabismus (exotropia or esotropia), amblyopia, glaucoma, macular degeneration, cataract, retinal detachment or nystagmus, or abnormality of the central cornea, lens, iris, ciliary body, or central retina. -
8. Presence of any medical condition predisposing the subject to craniofacial anomalies, degenerative myopia, or abnormal ocular refractive anatomy (e.g., osteogenesis imperfecta or Stickler, Down, Ehlers-Danlos, Donnai-Barrow, Treacher-Collins, or Apert/Crouzon/ Pfeiffer syndrome). -
9. Active or recent (within 2 weeks prior to screening) bacterial, viral, or allergic conjunctivitis. -
10. Active allergies causing uncontrolled ocular and nasal symptoms. -
11. Active sinusitis. -
12. Current or previous hypothyroidism or hyperthyroidism. -
13. Ongoing or recent (within 3 months prior to screening) chronic use of eyedrops containing preservatives such as benzalkonium chloride (BAK), Purite, or Polyquad. -
14. History of uncontrolled gastroenteric reflux disease or deviated nasal septum. -
15. If a female of childbearing potential (FOCBP):

    1. Are pregnant or lactating.
    2. Are unwilling to use an effective form of contraception (e.g., hormonal, oral, transdermal, implant, injection, or abstinence) for the duration of the study. -
16. A male subject with a partner who is a FOCBP unwilling to use an effective form of contraceptives (e.g., barrier, hormonal, oral, transdermal, implant, injection, or abstinence) for either themselves or their partner, as appropriate, for the duration of the study. -

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-02-04 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | From enrollment to the end of treatment at 6 weeks
  Change from baseline in corrected distance visual acuity (CDVA) with Early Treatment Diabetic Retinopathy Study (ETDRS) in the study eye (SE) at all post-baseline visits. The change in ETDRS scores will be recorded as logMAR scores and letters missed on the eye chart. A logMAR of 0.0 corresponds to 20/20 vision; higher values indicate greater myopia (near-sighted), and lower values indicate greater hyperopia (far-sighted) .
Change in eye assessments | From enrollment to the end of treatment at 6 weeks
  Clinically significant Abnormalities in ocular assessments at any post-baseline visit
Punctal stenosis or Bloody discharge | From enrollment to the end of treatment at 6 weeks
  Development of punctal stenosis or bloody discharge over the course of the study
Change in ocular assessments | From enrollment to the end of treatment at 6 weeks
  Change from baseline in ocular symptoms assessment (discomfort, burning, irritation, photophobia, and redness) at all post-baseline visits.

CONTACTS AND LOCATIONS:
Locations (1):
- Total Eye Care, P.A., Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified patient data that underlie the results reported in future publications, along with the protocol and statistical analysis plan, will be made available upon reasonable request. Data will be available beginning 12 months following publication and may be accessed by qualified researchers who submit methodologically sound proposal, subject to approval and execution of a data sharing agreement